CLINICAL TRIAL: NCT03403491
Title: Pilot-scale, Randomized Study Comparing Self-monitoring of Weight and Blood Pressure Via an Electronic Health Journal (patientMpower Platform) With Usual Care in Haemodialysis Patients
Brief Title: Study of Self-monitoring of Weight & Blood Pressure (Via patientMpower Platform) in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: patientMpower Ltd. (Industry)
Collaborators: Health Service Executive, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Hemodialysis patientMpower02
Record Dates: First submitted 2018-01-05; First posted 2018-01-18 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Renal Dialysis

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, sham-controlled, observational study. Usual care run-in period (2 weeks) followed by random order 2 x 4-week crossover periods. Comparison is active pMp app [+ digital weighing scales + BP monitor] for 4 weeks vs. sham application for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): Usual care for 2 weeks followed by using patientMpower application [+digital weighing scales & BP monitor] for 4 weeks followed by sham application (without digital scales or BP monitor) for 4 weeks.
  Interventions: Other: patientMpower application; Other: sham application
- Sequence 2 (Other): Usual care for 2 weeks followed by sham application (without digital scales or BP monitor) for 4 weeks followed by using patientMpower application [+digital weighing scales & BP monitor] for 4 weeks.
  Interventions: Other: patientMpower application; Other: sham application

INTERVENTIONS:
Other: patientMpower application — electronic health journal for patient to record weight, blood pressure, medication adherence and symptoms
Other: sham application — dummy application which does not allow recording of weight, blood pressure, medication adherence and symptoms

SUMMARY:
Pilot-scale study to assess the effect of self-monitoring using the patientMpower electronic health journal (pMp app) [+digital weighing scales & BP monitor] on outcomes in ambulatory haemodialysis patients. Design: prospective, open-label, random order, sham-controlled, two-period crossover comparison of the pMp app [+digital weighing scales & BP monitor] compared with a sham application (without weighing scales or BP monitor). Duration: 10 weeks (usual care run-in for 2 weeks followed by 2 x 4 observation periods).

Primary objective is to determine the frequency of use of the pMp app [+digital weighing scales & BP monitor] in patients randomized to that observation method. Additional objectives are to determine the effect of pMp app [+digital weighing scales & BP monitor] on proportion of haemodialysis sessions in which ultrafiltration rate is ≤ 10 mL/kg/h and in which interdialytic weight gain (IDWG) is ≤ 4% and effect of pMp on pre-dialysis weight and BP, medication adherence, compliance with daily recording (of fluid intake, weight, BP) and requirement for additional unscheduled dialysis.

An additional objective is to assess the acceptability and utility of the pMp app in helping hemodialysis patients and their healthcare professional caregivers manage their condition (assessed from both patient and healthcare professional perspective).

DETAILED DESCRIPTION:
Pilot-scale, prospective, open-label, randomized, two-period, cross-over intervention study.

Each patient will be randomized to one of the two possible observation sequences:

Sequence 1: run-in (2 weeks): usual care followed by period 1 (4 weeks): patientMpower application (+digital weighing scales & BP monitor) followed by period 2 (4 weeks): sham application

OR

Sequence 2: run-in (2 weeks): followed by period 1 (4 weeks) sham application followed by period 2 (4 weeks): patientMpower application (+digital weighing scales & BP monitor)

The study will not make any other changes to the therapeutic interventions offered to the patients. Patients will follow their usual care and hemodialysis programme throughout the study.

Proposed sample size is approximately 50 patients.

Patients will be recruited through three haemodialysis facilities under the governance of Beaumont Hospital, a tertiary care centre for nephrology in Dublin, Ireland.

The study observational intervention is an electronic health journal, the patientMpower application (with a supplied digital weighing scales and BP monitor). This has been developed specifically for patients undergoing hemodialysis. The app is an electronic application downloaded to the patient's mobile phone or tablet device. The app is designed to allow the patient to report various parameters relevant to hemodialysis and record these on a regular basis, ideally daily. The information recorded by the patients will be stored in a secure cloud system and will be available to the patient through their phone or mobile device at all times. No personal health data are stored on the phone or mobile device itself.

Patient-reported measures (at a minimum) will include body weight (at least one reading /day), BP and compliance with relevant medication. Additional patient-reported measures which can be reported on the patientMpower app include body temperature, activity levels and symptoms.

The control observation will be usual care with a sham electronic application (which will not allow recording of body weight, BP or other measurements).

The objective of this pilot-scale cross-over open label randomized study is to assess the effect of self-monitoring using the patientMpower electronic health journal [+digital weighing scales &BP monitor] on outcomes in ambulatory hemodialysis patients.The primary objective will be to determine the frequency of use of the patientMpower app (+digital weighing scales & BP monitor).

ELIGIBILITY:
Inclusion criteria:

* Requires maintenance hemodialysis in an ambulatory care setting.
* Aged at least 18 years.
* Has daily unrestricted access to a suitable smart phone or tablet device at home.
* Has an e-mail address.
* Has home broadband and/or mobile data as part of their mobile phone service.
* Demonstrates understanding of correct use of the patientMpower application, digital weighing scales, BP monitor and other study equipment.
* Capable and willing to perform measurements (e.g. weight, BP) at home and record information on the patientMpower application on a daily basis.
* Willing to give written informed consent.

Exclusion Criteria:

* Significant confusion or any concomitant medical condition, which would limit the ability of the patient to record symptoms or other parameters on an electronic health journal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renal Dialysis Centre, Principal Investigator — Beaumont Hospital, Dublin 9, Ireland
Locations (1):
- Renal Dialysis Centre, Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandys V, Bhat L, O'Hare E, Hudson A, O'Seaghdha CM, Sexton DJ. Interpretability of Home Blood Pressure Measurements in Haemodialysis A Post Hoc Analysis of a Randomised Cross-Over Study. Nephrology (Carlton). 2025 Sep;30(9):e70112. doi: 10.1111/nep.70112. PMID 40854574

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started | 20 | 23
Completed (Definition: at least 21 days of patient-reported weight data) | 17 | 18
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Population: All randomised patients who started the study observations
Groups:
- All Patients: All patients who started patientMpower observation period
Arm/Group | All Patients
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.42 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 39
  black | 3
  Asian | 1
Region of Enrollment [Number; unit: participants]
  Ireland | 43
time since first-ever hemodialysis [Mean (Standard Deviation); unit: years] | 3.44 (3.71)
vascular access modality [Count of Participants; unit: Participants]
  permcath | 25
  arteriovenous fistula | 18

OUTCOME MEASURES:

1. Primary Outcome: Patient Engagement With patientMpower App to Record Body Weight
Description: Actual number of days body weight reported by patient on patientMpower app
Time Frame: 28 days
Population: All patients who started patientMpower observation period and who recorded weight at least once
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 43
days | 24 (6)

2. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Ultrafiltration Rate (Proportion </= 10mL/kg/h)
Description: Proportion of hemodialysis sessions in which ultrafiltration rate is less than/equals 10mL/kg/h
Time Frame: 28 days
Population: Average of the proportion of hemodialysis sessions per patient in which ultrafiltration rate is less than/equals 10 mL/kg/h in observation period
Measure: Median (Inter-Quartile Range); unit: proportion of sessions
Groups:
- Sham: sham observation period
- patientMpower: patientMpower observation period
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
proportion of sessions | 0.83 [0.25 to 1.00] | 0.83 [0.44 to 1.00]

3. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Interdialytic Weight Gain (Relative to Dry Weight)
Description: Average interdialytic weight gain as percentage of patient's dry weight
Time Frame: 28 days
Population: Average of interdialytic weight gain per patient for all haemodialysis sessions in each observation period
Measure: Mean (Standard Deviation); unit: % of dry weight
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
% of dry weight | 2.76 (0.96) | 2.68 (0.92)

4. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Interdialytic Weight Gain (Absolute)
Description: Average interdialytic weight gain in kg
Time Frame: 28 days
Population: Average of interdialytic weight gain per patient for all haemodialysis sessions in each observation period
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
kg | 2.29 (0.74) | 2.22 (0.71)

5. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Interdialytic Weight Gain (Proportion </= 4%)
Description: Proportion of hemodialysis sessions in which interdialytic weight gain is less than/equals 4%
Time Frame: 28 days
Population: Average of the proportion of hemodialysis sessions per patient in which interdialytic weight gain is less than/equals 4% in observation period
Measure: Median (Inter-Quartile Range); unit: proportion of sessions
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
proportion of sessions | 0.83 [0.67 to 1.00] | 0.83 [0.67 to 1.00]

6. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Predialysis Weight
Description: predialysis weight
Time Frame: 28 days
Population: average of the pre-dialysis clinic observed weights per patient in the observation period
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
kg | 89.15 (23.30) | 89.27 (23.34)

7. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Pre-dialysis Systolic Blood Pressure
Description: pre-dialysis supine systolic blood pressure
Time Frame: 28 days
Population: average of the clinic-observed pre-dialysis supine systolic blood pressures per patient in the observation period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
mmHg | 146.6 (18.4) | 146.3 (19.6)

8. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Pre-dialysis Diastolic Blood Pressure
Description: pre-dialysis supine diastolic blood pressure
Time Frame: 28 days
Population: average of the clinic-observed pre-dialysis supine diastolic blood pressures per patient in the observation period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 41 | 41
mmHg | 75.2 (14.8) | 74.5 (15.2)

9. Secondary Outcome: Patient Engagement With patientMpower App to Record Medication Adherence
Description: actual number of days medication adherence reported by patient on patientMpower app
Time Frame: 28 days
Population: All patients who started patientMpower observation period and recorded medicines adherence at least once
Measure: Mean (Full Range); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 2
days | 18 [16 to 21]

10. Secondary Outcome: Patient Engagement With patientMpower App to Record Blood Pressure.
Description: actual number of days blood pressure reported by patient on patientMpower app
Time Frame: 28 days
Population: All patients who started patientMpower observation period and who recorded blood pressure at least once
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 38
days | 18 (8)

11. Secondary Outcome: Patient Engagement With patientMpower App to Record Symptoms
Description: Actual number of days symptoms reported by patient on patientMpower application
Time Frame: 28 days
Population: All patients who started patientMpower observation period and who recorded symptoms at least once on patientMpower app
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 33
days | 13 (8)

12. Secondary Outcome: Patient Engagement With patientMpower App to Record Fluid Intake
Description: Actual number of days fluid intake reported by patients on patientMpower application
Time Frame: 28 days
Population: All patients who started patientMpower observation period and who recorded fluid intake at least once on patientMpower app
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 33
days | 13 (8)

13. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Requirement for Additional Unscheduled Hemodialysis.
Description: number of patients requiring additional unscheduled hemodialysis sessions
Time Frame: 28 days
Population: All patients who started the sham or patientMpower observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 43 | 43
Participants | 2 | 2

14. Secondary Outcome: Patient Opinion on Utility and Acceptability of patientMpower Application
Description: Questionnaire-based assessment: 7 questions. [pMp = patientMpower intervention]
  1. using pMp helped me to take correct dose of my medicines every day
  2. using pMp gave me more confidence/greater sense of control in managing my health
  3. my preference for using pMp
  4. my difficulty rating in using pMp
  5. effect of using pMp on my well-being and daily life
  6. do I want to continue using pMp after study end
  7. did I like using pMp Possible responses Q1, Q2: strongly agree/agree/disagree/strongly disagree; Q3: yes/no preference/no; Q4: very easy/easy/difficult/very difficult; Q5: positive/negative; Q6: yes/no; Q7: 10-point linear scale: 1 (did not like at all) to 10 (liked a lot)
Time Frame: 28 days
Population: All patients who started the patientMpower observation period and provided a response to the questionnaire
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 23
participants
  pMp helped me take my correct medicines/day | 12
  pMp gave me greater confidence/control | 19
  preferred using pMp = yes | 14
  pMp easy or very easy to use | 21
  positive effect pMp on well-being/daily life = yes | 19
  want to continue using pMp after study end = yes | 18
  liked using pMp: score at least 8/10 | 15

15. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Pre-dialysis Inferior Vena Cava Collapsibility
Description: number of patients with at least 50% collapsibility
Time Frame: 28 days
Population: All patients who had measurement of inferior vena cava diameter assessed pre-dialysis
Measure: Count of Participants; unit: Participants
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 7 | 7
Participants | 7 | 6

16. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Pre-dialysis Inferior Vena Cava Longitudinal Diameter
Description: longitudinal diameter
Time Frame: 28 days
Population: All patients who had measurement of inferior vena cava diameter assessed pre-dialysis
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 7 | 7
cm | 1.7 (0.5) | 1.8 (0.5)

17. Secondary Outcome: Effect of patientMpower App [+Digital Scales & BP Monitor] on Pre-dialysis Inferior Vena Cava Transverse Diameter
Description: transverse diameter
Time Frame: 28 days
Population: All patients who had measurement of inferior vena cava diameter assessed pre-dialysis
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Sham | patientMpower
Number analyzed (Participants) | 7 | 7
cm | 1.5 (0.6) | 1.5 (0.6)

ADVERSE EVENTS:
Time Frame: Observation duration for sham observation period = 28 days for all patients who started sham observation period. Observation duration for patientMpower observation period = 28 days for all patients who started patientMpower observation period. Design was randomised 2 x 28 day crossover
Groups:
- Sham Observation Period: All patients who started sham observation period
- patientMpower Observation Period: All patient who started patientMpower observation period
Arm/Group | Sham Observation Period | patientMpower Observation Period
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/43
Other Adverse Events (participants affected / at risk) | 0/43 | 1/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Observation Period (N=43) | patientMpower Observation Period (N=43)
leg fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1) — alcohol withdrawal seizure reported in same patient
alcohol withdrawal seizure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — hypertension reported in same patient
arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Observation Period (N=43) | patientMpower Observation Period (N=43)
fall (General disorders) | 0 (0) | 1 (2) — fell off weighing scales twice

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03403491/Prot_000.pdf
  • Statistical Analysis Plan: Description (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03403491/SAP_001.pdf
  • Statistical Analysis Plan: Appendix 1 (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03403491/SAP_002.pdf